CLINICAL TRIAL: NCT00774605
Title: A Phase 1, Open-Label, Nonrandomized, Single Dose Study To Characterize The Pharmacokinetics Of A Varenicline (CP-526,555) Transdermal Solution And A Varenicline Transdermal Delivery System Applied To The Skin Of Adult Smokers
Brief Title: A Study Evaluating The Absorption Of Varenicline Into The Body From A Varenicline Solution And A Varenicline Patch Applied To The Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: A3051118
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Smoking Cessation
Keywords: percutaneous, transcutaneous, topical, varenicline, transdermal, transdermal delivery system, patch
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline free base solution (Experimental)
  Interventions: Drug: Varenicline free base solution
- Varenicline transdermal delivery system (Experimental)
  Interventions: Drug: Varenicline free base patch

INTERVENTIONS:
Drug: Varenicline free base solution — A single application of a 4.8 mg varenicline solution will be applied to the upper back over a 24 hour period
  Arms: Varenicline free base solution
Drug: Varenicline free base patch — A single application of a nominal 1.2 mg dose of a varenicline transdermal delivery system (5 cm2 patch, 4.8 mg drug payload) will be applied to the upper back over a 24 hour period
  Arms: Varenicline transdermal delivery system

SUMMARY:
To evaluate the absorption, safety, and tolerability of a varenicline solution and a varenicline patch applied to the skin.

DETAILED DESCRIPTION:
Additional Study Purpose Details: Evaluation of the pharmacokinetic profile of a varenicline solution and a varenicline patch applied to the skin

ELIGIBILITY:
Inclusion Criteria:

* healthy, adult, male smokers

Exclusion Criteria:

* significant medical illness

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Varenicline area under the curve from 0 to the last quantifiable concentration (AUClast) and varenicline area under the curve from 0 to infinity (AUCinf) | 8 days

SECONDARY OUTCOMES:
Evaluation of adverse events (including skin irritation) | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051118&StudyName=A%20Study%20Evaluating%20The%20Absorption%20Of%20Varenicline%20Into%20The%20Body%20From%20A%20Varenicline%20Solution%20And%20A%20Varenicline%20Patch%20Applied%20To%20The%20Sk